CLINICAL TRIAL: NCT05083000
Title: Phase I Dose-escalation Study of Topotecan in Moderate-severe COVID-19 Patients
Brief Title: Reducing Hypoxia in Patients With Coronavirus Disease (COVID-19) Using Topotecan With Standard of Care
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Christian Medical College, Vellore, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TOTORO1
Record Dates: First submitted 2021-10-11; First posted 2021-10-19 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-09

CONDITIONS: COVID-19 Respiratory Infection
Keywords: Topotecan; hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Topotecan

STUDY DESIGN:
Intervention Model Description: The dose escalation will be in a standard 3+3 dose escalation design with 0.25mg increments of Topotecan; it will begin with a single dose 0.25mg for 3 patients-expanded to another 3 if no toxicities are seen. Subsequent dose levels will be 2 doses of 0.25mg, a single dose of 0.5mg and then 2 doses of 0.5mg (maximum of 24 patients).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topotecan (Experimental): Subject will receive Topotecan as a single dose or 2 consecutive doses given via intravenous (IV). The starting dose level of Topotecan is 0.25mg. Subsequent dose levels will be 2 doses of 0.25mg, a single dose of 0.5mg and then 2 doses of 0.5mg.
  Standard of care treatments for COVID-19 will be given together if available as per the following protocol:
  1. IV Dexamethasone 6mg once daily for at least 5 days and not more than 10 days.
  2. IV Remdesivir 200mg loading dose on day 1 followed by 100mg once daily for 4 days.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Topotecan — Topotecan hydrochloride is a semi-synthetic derivative of camptothecin and is an anti-tumor drug with topoisomerase I-inhibitor activity. It is a well-established chemotherapeutic agent used for cancer treatment.
  Other Names: Topotecan hydrochloride

SUMMARY:
The primary objective of the phase 1 trial is to identify a dose of topotecan that will be safe to take forward into a Phase 2 trial, with no unexpected toxicities or drug-drug interactions with standard therapy for COVID-19. The investigators hypothesise that a single dose of low-dose Topotecan will blunt the expression of inflammatory genes in patients with moderate COVID-19, without cytotoxic side effects.

DETAILED DESCRIPTION:
4 fixed dosing levels (0.25 -0.5mg) of Topotecan will be evaluated in this trial, using sub-cytotoxic doses of Topotecan which are well below typical chemotherapy levels and shown not to cause myelosuppression in previously tested populations. The dose escalation will be in a standard 3+3 dose escalation design with 0.25 mg increments of Topotecan. The study aims to establish the recommended phase 2 dose (RP2D) of Topotecan in hypoxic patients with moderate to severe COVID-19.The RP2D is defined as the maximum safe dose at which 3 or more patients are found to have clinically relevant concentrations of Topotecan in the blood stream, without reaching anti-cancer concentrations in plasma (defined as Area under the curve (AUC)>150000) and without causing Grade 2/3/4 neutropenia (CTCAE5).

ELIGIBILITY:
Inclusion Criteria:

* Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection confirmed by at least 1 positive Polymerase Chain Reaction (PCR) test
* Moderate COVID as evidenced by Oxygen saturation <93% on room air (or <88% if prior CLD)
* Admission to emergency department for monitoring and/or supportive care:
* The following biochemical markers:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L. Platelets ≥ 100 x 109/L, Haemoglobin ≥ 9x 109/L.
* Bilirubin < 1.5 times upper limit of normal (ULN). Alanine aminotransferase (ALT) and Aspartate Aminotransferase (AST) < 2.5 times ULN.
* Calculated creatinine clearance of ≥ 30ml/min calculated using the formula of Cockcroft and Gault: (140-age) x mass (kg)/)72x creatinine mg/dl); multiple by 0.85 if female.
* Laboratory features of cytokine release, as defined by any 1 of the following:

  i. C-reactive protein (CRP)> 75mg/L ii. Lactate Dehydrogenase (LDH) > ULN iii. D-dimer > 1.0 mg/L iv. Ferritin > 500ng/ml v. Elevated Interleukin-6 levels

Exclusion Criteria:

* Patients requiring mechanical ventilation
* Any immunosuppressive medication including chemotherapy(excluding steroids) administered concurrently or within last 14 days.
* Patients with uncontrolled diabetes mellitus (HbA1C within 1 month >8)
* Pregnancy or Breastfeeding.
* Known allergy to Topotecan. Unconjugated hyperbilirubinemia on a fasting Liver Function Test (LFT), which can indicate Gilberts Syndrome.
* Suspected active bacterial, fungal, or other infection in addition to COVID-19.
* Any condition that would, in the opinion of the Investigator, increase the risk of the participant
* by participating in the study.
* Inability to provide consent.
* Unable to comply with study procedures.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerable dose of Topotecan | 24 hours and 14 days from the time of Topotecan administration
  To determine a maximal dose of Topotecan, at which less than 1 out of 3 patients exhibit anti-cancer concentrations in plasma, or have G2/3/4 neutropenia

SECONDARY OUTCOMES:
Rate of reduction in the duration of supplemental oxygen requirement in participants | 1 week from administration of Topotecan
  Determine effect of Topotecan on duration of additional oxygen requirements
Rate of treatment related CTCAE grade 3/4 haematological toxicity | Up to Day 10 from Topotecan administration
  Dose limiting toxicities will be graded using CTCAE version 5.0.
Number of participant with Serious Adverse Events | Within 14 days from Topotecan administration
  Serious Adverse Events experience by subject after Topotecan administration (related and unrelated).
Proportion of patients requiring ICU care | 28 days from Topotecan administration
  Number of patients requiring intubation/inotropic/vasopressor support
Proportion of patients requiring mechanical ventilation | 28 days from Topotecan administration
  Number of patients requiring mechanical ventilation
Time to discharge | 28 days from Topotecan administration
  Time to hospital discharge in days
Proportion of patients with secondary infections | 28 days from Topotecan administration
  Number of patients with secondary infections
Proportion of patients who died after enrolment into trial | 28 days from Topotecan administration
  Death from related and unrelated causes

CONTACTS AND LOCATIONS:
Overall Officials: Anand JEYASEKHARAN, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No